CLINICAL TRIAL: NCT02879916
Title: Comparison of the Analgesic Effect of Levobupivacaine 0.5% Via Interscalene Nerve Block or Via Interscalene Nerve Block Combined With a Stellate Ganglion Block in Patients Undergoing Shoulder Arthroscopy With General Anaesthesia
Brief Title: Comparison of an Interscalene Nerve Block With or Without Stellate Ganglion Block for Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, research assistant, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/20/162; B300201111454 (Registry Identifier: FAGG)
Record Dates: First submitted 2016-08-11; First posted 2016-08-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia, Regional
MeSH Terms: interventions — Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): NaCl 0.9% 3ml perineural stellate ganglion injection
  Interventions: Drug: NaCl 0.9%
- Stellate ganglion block (Active Comparator): Levobupivacaine 3ml perineural stellate ganglion injection
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Inject 3ml of levobupavacaine into the stellate ganglion area
  Arms: Stellate ganglion block
Drug: NaCl 0.9% — Inject 3ml of NaCl 0.9% into the stellate ganglion area
  Arms: Placebo

SUMMARY:
This study describes the difference of analgesic effect of levobupivacaine 0.5% administered through an interscalene nerve block with or without a stellate ganglion block. The length of the analgesic effect is our primary outcome parameter. Half of the recruited patients will receive a stellate ganglion block and half of the patients won't.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 to 3
* Need for shoulder surgery

Exclusion Criteria:

* Mental retardation
* allergy for local anesthetics
* a medical reason as a contra-indication for NSAID use
* Diabetes mellitus
* peripheral neuropathy
* chronic analgetic use
* chronic pain patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  The duration of analgesia assessed with quantitative sensory testing

SECONDARY OUTCOMES:
Need for rescue analgesia | 24 hours
  The timing of the need for rescue analgesia as requested by the patient
Duration of motor block | 24 hours
  The duration of a motor block

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sermeus, MD, Principal Investigator — Consultant

IPD SHARING:
Plan to Share IPD: No